CLINICAL TRIAL: NCT03466892
Title: RTFM-AB - Repetitive Thinking in FibroMyalgia and Attentional Bias: Links Between Attentional Bias in Later Stages of Attention and Tendency to Repetitive Thinking
Brief Title: Repetitive Thinking in FibroMyalgia and Attentional Bias
Acronym: PRFM-BA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0003
Record Dates: First submitted 2018-02-28; First posted 2018-03-15 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
Keywords: Repetitive Negative Thinking; Rumination; Fibromyalgia; Chronic pain; Attentional Bias
MeSH Terms: conditions — Chronic Pain; Rumination Syndrome; Fibromyalgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires and computer paradigm — Patients will complete different scales and also the visual probe task. First, we hypothesize the attention bias for pain-related information in the FM group is correlated with the level of negative repetitive thinking in the maintained attention phase. Second, we hypothesize the attention bias is more important in the attention maintenance phase (1250 ms) than in the attention orientation phase (500 ms).

SUMMARY:
Theoretical models of chronic pain hypothesize a privileged treatment of pain-related information that would be the basis of avoidance behaviors in chronic pain. This privileged treatment, also called attentional bias, has been found experimentally in chronic pain. Meta-analyses confirmed that but leaded the question of the difference found between bias in period of attention orientation and bias in period of maintained attention. One of the hypotheses is to consider one or more cognitive processes that would "fix" the attention around significant perceived problems and that would hinder the attentional disengagement and the reorientation of attention towards neutral or positive stimuli. In view of the scientific literature in psychopathology but also in chronic pain we think that the negative repetitive thoughts (RNT) variable is one of these processes. So the investigators want to better understand the difference of attentional bias at different moments of the attentional process by interrogating the Repetitive Thinking variable. More specifically the investigators test the Attentional Bias hypothesis in Fibromyalgia. Patient with Fibromyalgia will be recruited at the Pain Center of CHU-Amiens. Patients will complete different scales and also the visual probe task. First, the investigators hypothesize the attention bias for pain-related information in the FM group is correlated with the level of negative repetitive thinking in the maintained attention phase. Second, the investigators hypothesize the attention bias is more important in the attention maintenance phase (1250 ms) than in the attention orientation phase (500 ms).

ELIGIBILITY:
Inclusion Criteria:

Adults Patients inclusion criteria:

* 1990 ACR Criteria of FM
* Free and informed consent signed.
* French mother tongue spoken, written, read.
* Major person.

Exclusion Criteria:

* Adult major under protection.
* Patient with severe psychosis or depression or severe anxiety or impulsivity as -assessed by the clinician.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: One group. It is a cross sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
To measure attentional bias using a visual probe task paradigm. | 1 hour and 20 min

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: Undecided